CLINICAL TRIAL: NCT06476574
Title: Retentive Capacity of Bonded Retainer Versus Vacuum-formed and Combined Bonded-vacuum Retainers: A Randomized Controlled Clinical Trial
Brief Title: Retentive Capacity of Bonded Retainer Vs Vacuum-formed and Combined Bonded-vacuum Retainers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Ayman Ahmed El Behery, Master Degree student, Orthodontics department, Faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: derosuperstar123
Record Dates: First submitted 2024-05-14; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Orthodontic Retainer; Fixed Orthodontic Retainer; Orthodontic Relapse; Essix Retainer; Vacuum-formed Retainer; Dual Retention Protocol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vacuum-formed retainer (Experimental): An alginate impression will be taken to be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used.
  Interventions: Device: Vacuum-formed retainer
- Combined Vacuum-formed and Lingual bonded retainer from canine-to-canine. (Experimental): A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors; followed by an alginate impression; the impression will be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used.
  Interventions: Device: Combined Vacuum-formed and Lingual bonded retainer from canine-to-canine.
- Lingual bonded retainer from canine-to-canine (Active Comparator): A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors.
  Interventions: Device: Lingual bonded retainer from canine-to-canine

INTERVENTIONS:
Device: Vacuum-formed retainer — * After patient finishes orthodontic treatment, the fixed orthodontic appliance will be debonded; finishing and polishing of the enamel surface will be done.
  * An alginate impression will be taken to be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used.
  * The retainer will be finished and delivered to the patient.
  * The patient will be instructed to wear the retainer night time only and to contact us if any damage occurred to the retainers for immediate replacement; and he will be supplied with a check list to evaluate the compliance and to calculate the wearing hours.
  * Another alginate impression will be taken for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0 (before wearing of the retainer).
  Arms: Vacuum-formed retainer
Device: Combined Vacuum-formed and Lingual bonded retainer from canine-to-canine. — * A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors; followed by an alginate impression; the impression will be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used & it will be finished and delivered to the patient.
  * The patient will be instructed to wear the Vacuum retainer night time only and to contact us if any damage occurred to the retainers for immediate replacement or rebonding of the detached parts of the bonded retainer; and will be supplied with a check list to evaluate the compliance and to calculate the wearing hours.
  * Another alginate impression will be taken (with the bonded retainer in place) for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0.
  Arms: Combined Vacuum-formed and Lingual bonded retainer from canine-to-canine.
Device: Lingual bonded retainer from canine-to-canine — * After patient finishes orthodontic treatment, the fixed orthodontic appliance will be debonded; finishing and polishing of the enamel surface will be done.
  * A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors.
  * The patient will be instructed to contact us if any damage occurred to the retainers for immediate replacement or rebonding of the detached parts of the retainer.
  * An alginate impression will be taken (with the bonded retainer in place) for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0 (at the same visit of the delivery of the bonded retainer).
  Arms: Lingual bonded retainer from canine-to-canine

SUMMARY:
The main goal is to test the differences between the retentive capacity of fixed retainer, vacuum-formed retainer & combination of both; and recommend the most effective protocol for retention of lower incisors crowding treated by non-extraction treatment plan

The main question is: In patients with lower incisors crowding treated by non-extraction treatment plans, what is the difference in retentive capacity between fixed retainer, vacuum formed retainer and combined bonded and vacuum retainers in maintaining corrected lower anterior segment crowding? After enrolment, each participant will have the orthodontic appliance debonded, the adhesive remnant removed and the enamel surface polished. An alginate impression will be taken to be poured into a study model which will be scanned to obtain STL files for digital models. All patients will have periodontal charting and probing depths recorded for the lower anterior segment. According to the randomization, each patient will be assigned to a group to receive the retainer. All patients will be called for follow-up after 1 week, 1 and 3 months.

DETAILED DESCRIPTION:
Research objective: Retention is a key part of success of orthodontic treatment. Unless we can maintain the teeth in position after orthodontic treatment, the beneficial results of the treatment can be lost. There are currently many different types, designs and materials of removable and fixed retainers and it is unclear which retainers are the best, and how long they should be used for. There is also little knowledge about the possible adverse effects on the Periodontal health, patients' satisfaction and compliance are better with which type of retainers; and which retainers have the greatest failure rate. The dual retention protocol -combined vacuum and fixed retainers- is widely used among clinicians but without strong evidence on its effectiveness compared to the use of single retainer.

Research procedure in brief:

This study will be carried out on patients enrolled from the Outpatient Clinic of Orthodontics department, Faculty of Dentistry, Cairo University.

Eligibility criteria:

Inclusion criteria:

* Adult patients
* Finished non-extraction orthodontic treatment
* Full set of permanent dentition (excluding third molars).
* Good oral hygiene
* No restorations on lower anterior teeth or morphologic crown anomalies.
* Little's irregularity index score 0

Exclusion criteria:

* Systemic disease or drugs affecting periodontal health.
* Smokers
* Poor oral health that precludes orthodontic treatment (presence of caries, active white spots, or periodontal diseases).

Interventions:

* Every patient will be examined for any systemic disease or dental hard or soft tissue pathology, and the eligibility for previously mentioned eligibility criteria will be checked.
* The purpose of the study and the details of the intervention and control will be explained for the patient and they will be asked whether they are willing to
* participate in the study and accordingly will sign an informed consent. Post orthodontic treatment records (study models, digital models and intra-oral photos) will be taken for every patient as part of the routine procedure for the treatment of patients in the outpatient clinic of the Orthodontic Department, Cairo University. And used as pre-intervention records

Clinical Procedure:

* After taking post-treatment records, every patient will have the orthodontic appliance debonded, the adhesive remnant removed and the enamel surface polished
* An alginate impression will be taken to be poured into a study model.
* Study models will be scanned to obtain STL files for digital models.
* All patients will have periodontal charting and probing depth recorded for the lower anterior segment.
* According to the randomization, each patient will be assigned to a group to receive the retainer.
* All patients will be called for follow-up after 1 week, 1 and 3 months.

Intervention group I:

Vacuum-formed retainer.

* After patient finishes orthodontic treatment, the fixed orthodontic appliance will be debonded; finishing and polishing of the enamel surface will be done.
* An alginate impression will be taken to be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used.
* The retainer will be finished and delivered to the patient.
* The patient will be instructed to wear the retainer night time only and to contact us if any damage occurred to the retainers for immediate replacement; and he will be supplied with a check list to evaluate the compliance and to calculate the wearing hours.
* Another alginate impression will be taken for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0 (before wearing of the retainer).

Intervention group II:

Combined Vacuum-formed and Lingual bonded retainer from canine-to-canine.

* After patient finishes orthodontic treatment, the fixed orthodontic appliance will be debonded; finishing and polishing of the enamel surface will be done.
* A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors; followed by an alginate impression; the impression will be poured into a working model for fabrication of the Vacuum-formed retainer; 1mm Hard vacuum sheet will be used.
* The retainer will be finished and delivered to the patient.
* The patient will be instructed to wear the Vacuum retainer night time only and to contact us if any damage occurred to the retainers for immediate replacement or rebonding of the detached parts of the bonded retainer; and will be supplied with a check list to evaluate the compliance and to calculate the wearing hours.
* Another alginate impression will be taken (with the bonded retainer in place) for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0 (at the same visit of the delivery of the bonded retainer).

Control group III:

Lingual bonded retainer from canine-to-canine.

* After patient finishes orthodontic treatment, the fixed orthodontic appliance will be debonded; finishing and polishing of the enamel surface will be done.
* A multistrand rectangular stainless steel retainer wire will be bonded to the lingual surface of the lower anterior teeth, from the canine-to-canine bonded to all six anteriors.
* The patient will be instructed to contact us if any damage occurred to the retainers for immediate replacement or rebonding of the detached parts of the retainer.
* An alginate impression will be taken (with the bonded retainer in place) for fabrication of the study model which will later be scanned to obtain the digital model at T0; and a periodontal chart will be filled to record the periodontal status at T0 (at the same visit of the delivery of the bonded retainer).

All the three groups will be called for follow up after 1week T1, 1month T2 and 3 months T3.

At each follow up visit, an alginate impression will be taken to obtain a study cast which will be later scanned to get a digital model and a periodontal chart will be filled to evaluate the periodontal condition; also, the integrity of the retainers will be checked together with the rate of failure or debonding of the fixed retainer which will be recorded.

The compliance chart will be collected and a new one will be supplied.

Outcomes: Relapse, Patient's compliance and satisfaction, Periodontal health, Integrity of the retainer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Finished non-extraction orthodontic treatment
* Full set of permanent dentition (excluding third molars).
* Good oral hygiene
* No restorations on lower anterior teeth or morphologic crown anomalies.
* Little's irregularity index score 0

Exclusion Criteria:

* Systemic disease or drugs affecting periodontal health.
* Smokers
* Poor oral health that precludes orthodontic treatment (presence of caries, active white spots,or periodontal diseases)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
The stability of the orthodontic treatment result and the degree of relapse from baseline to 6 months | Relapse will be measured at 1 week, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  The stability of the orthodontic treatment result and the degree of relapse will be measured by superimposition of the digital model at each time point on the initial model after debonding at T0.

SECONDARY OUTCOMES:
Patient's compliance | It will be measured at 1 week, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  patients' compliance will be evaluated by the check list supplied at each time point for the groups using removable retainers.
Periodontal health | It will be measured at 1 week, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  Periodontal health will be monitored by a filling a periodontal chart at each time point to check the probing depth, bleeding on probing and calculus formation on the lingual surface of lower anteriors.
The integrity of the retainers | It will be measured at 1 week, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  The integrity of the retainers will be evaluated based on the rate of fracture/ debonding and loss of the retainer.
Patient's satisfaction | It will be measured at 1 week, 1 month, 3 months and 6 months after the intervention during the follow-up period and will be done by a single calibrated examiner
  Patients' satisfaction will be evaluated at each follow up visit, the patients in all groups will fill a questionnaire form.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer A. ElBehery, Bachelor, Principal Investigator — Cairo University; Fady H. Fahim, Ass Professor, Study Director — Cairo University; Sally M. Reyad, Lecturer, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt